CLINICAL TRIAL: NCT00524927
Title: A Phase IV, Randomized, Double Blind, Single Centre, Placebo Controlled Study to Assess the Safety and Efficacy of Methoxyflurane [Penthrox] for the Treatment of Incident Pain in Participants Undergoing a Bone Marrow Biopsy Procedure
Brief Title: Safety and Efficacy of Methoxyflurane for Treatment of Incident Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Developments International Limited (Industry)
Collaborators: Australian Department of Industry, Tourism and Resources (Industry)
Responsible Party: Greg Plunkett, Regulatory Affairs Manager, Medical Developments International
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06/61
Record Dates: First submitted 2007-09-02; First posted 2007-09-05 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Pain Measurement
Keywords: Incident Pain; Bone Marrow Biopsy
MeSH Terms: interventions — Methoxyflurane; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Methoxyflurane
- B (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Methoxyflurane
  Arms: A
Drug: Normal Saline
  Arms: B

SUMMARY:
This study aims to provide further supportive evidence that Methoxyflurane, a potent analgesic, administered using the Penthrox Inhaler is safe and efficacious in adult participants, specifically those who experience incident pain associated with a planned bone marrow biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (18 years of age or older)
* Able to give written informed consent
* Anticipated episode(s) of incident pain related to planned BMB lasting no more than 30 minutes on average
* Anticipated life expectancy of at least 1 month

Pre-Exclusion Criteria:

* Subjects with a clinical condition that may, in the opinion of the investigator, impact on the subject's ability to participate in the study, or on the study results
* Participants who have had IV sedation/opioid on previous BMB and who wish to receive IV sedation/opioid on this occasion or who in the opinion of the BMB operator would be advised to receive IV sedation/opioid on this occasion
* Concomitant use of other investigational agents
* Concomitant use of nephrotoxic agents such as gentamicin
* Uncontrolled INR (>4)
* Personal or familial hypersensitivity to fluorinated anaesthetics
* Personal or familial malignant hyperthermia
* Respiratory rate of less than 10 per minute
* Has previously received methoxyflurane
* Known pre-existing renal or hepatic impairment
* Compromised Renal Function (creatinine ≥ 1.5 x ULNR)
* Compromised Liver Function (bilirubin ≥ 2.5 x ULNR)

Exclusion Criteria:

* Premedication with anxiolytic (e.g. midazolam, diazepam)
* Dosed with breakthrough dose of analgesic that may contribute to control of pain during the planned procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2007-09; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Determine where there is a difference in efficacy between Methoxyflurane and placebo for control of pain in participants undergoing a Bone Marrow Biopsy

SECONDARY OUTCOMES:
Determine the safety of Methoxyflurane

CONTACTS AND LOCATIONS:
Overall Officials: Odette Spruyt, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Spruyt O, Westerman D, Milner A, Bressel M, Wein S. A randomised, double-blind, placebo-controlled study to assess the safety and efficacy of methoxyflurane for procedural pain of a bone marrow biopsy. BMJ Support Palliat Care. 2014 Dec;4(4):342-8. doi: 10.1136/bmjspcare-2013-000447. Epub 2013 Jun 7. PMID 24644183